CLINICAL TRIAL: NCT00002298
Title: Long-Term Efficacy and Tolerance of Oral Ribavirin Compared to Placebo as a Preventative in Early Stages of Human Immunodeficiency Virus Infection - United States
Brief Title: The Safety and Effectiveness of Ribavirin in the Early Stages of HIV-Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: ICN Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 013A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-03

CONDITIONS: HIV Infections
Keywords: Ribavirin; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirin

SUMMARY:
The objective of this clinical trial is to determine whether long-term oral dosage of ribavirin delays development of symptomatic HIV disease in HIV antibody positive subjects who are completely asymptomatic (CDC classification group II), who have only the lymphadenopathy syndrome (CDC classification group III), or who have clinical symptoms but not severe HIV disease as defined by CDC classification, and whether the dosage regimen is safe and tolerable in these subjects.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acyclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* CDC classification group IV A (ARC).
* CDC classification group IV C-1 (AIDS) and IV C-2 (including Thrush or Herpes zoster during the past 2 years). Positive plasma p24 antigen.
* Unstable medical condition, including serious cardiovascular, renal, hepatic, neurologic, infectious, or oncologic condition even if unrelated to HIV infection.
* Splenectomy.

Concurrent Medication:

Excluded:

* Isoprinosine.

Patients with the following are excluded:

* Failure to give informed consent.
* CDC classification group IV A (ARC).
* CDC classification group IV C-1 (AIDS) and IV C-2 (including Thrush or Herpes zoster during the past 2 years).

Positive plasma p24 antigen.

* Unstable medical condition, including serious cardiovascular, renal, hepatic, neurologic, infectious, or oncologic condition even if unrelated to HIV infection.
* Splenectomy.

Prior Medication:

Excluded within 4 weeks of start of screening tests:

* Zidovudine.
* Other drug with scientifically accepted anti-HIV properties.
* Scientifically accepted immunostimulant treatment.
* Immunosuppressant.
* Myelosuppressant or other known toxic drugs.

HIV infection group II (CDC), asymptomatic HIV infection.

* HIV antibody positive by Western blot with antibodies to p24 band and GP160 band and/or GP41. Two positive tests during screening will be required. CDC HIV infection group II, asymptomatic HIV infection, as defined in Appendix A, or CDC HIV infection group III, persistent generalized lymphadenopathy (PGL, formerly LAS).
* OKT4+ lymphocyte count greater than 300 cells/mm3 and less than 600 cells/mm3. The counts will be determined on three separate evaluations separated by at least 7 days between evaluations. These three counts will be averaged and for inclusion in the study the mean of the OKT4+ lymphocyte count must be greater than 200 cells/mm3 and less than 600 cells/mm3. Conclusion of screening tests:
* Within 42 days of starting them. Patients must be entered into the study within 14 days of screening completion. Ability to participate as outpatient:
* Ambulatory, competent to sign informed consent, and able to cooperate with the treatment plan and evaluation schedule. Informed consent:
* Must be signed before randomization to treatment. Physical activity evaluation with Karnofsky score greater than or equal to 90.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult